CLINICAL TRIAL: NCT03462472
Title: The Acute Effects of Leg Heating and Transcutaneous Electrical Nerve Stimulation on Leg Blood Flow and Functional Capacity in Those With Peripheral Arterial Disease
Brief Title: Effect of Lower Leg Heating and Transcutaneous Electrical Nerve Stimulation on Exercise Capacity in Patients With PAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salisbury University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11112015-2
Record Dates: First submitted 2018-02-13; First posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 15 minute lower leg heating (Experimental)
  Interventions: Behavioral: Lower leg heating
- 45 minute lower leg heating (Experimental)
  Interventions: Behavioral: Lower leg heating
- Control (No Intervention)
- 15 minute lower leg TENS (Experimental)
  Interventions: Behavioral: Lower leg transcutaneous electrical nerve stimulation (TENS)
- 45 minute lower leg TENS (Experimental)
  Interventions: Behavioral: Lower leg transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Behavioral: Lower leg heating — Immersion of lower legs in a circulating water bath at a temperature of 42 degrees Celsius
  Arms: 15 minute lower leg heating; 45 minute lower leg heating
Behavioral: Lower leg transcutaneous electrical nerve stimulation (TENS) — Bilateral lower leg transcutaneous electrical nerve stimulation (TENS) using burst mode at a 3Hz burst rate, 100Hz frequency, and 250 µs pulse duration, sufficient to evoke skeletal muscle contraction
  Arms: 15 minute lower leg TENS; 45 minute lower leg TENS

SUMMARY:
Peripheral arterial disease (PAD) is characterized by poor circulation in the lower extremities that often provokes claudication (leg pain, numbness, and heaviness) with physical exertion. The aim of this research protocol is to determine the effect of two non-invasive treatment modalities on leg blood flow and exercise capacity in those with PAD. Specifically, we are measuring popliteal artery blood flow (Doppler ultrasound), toe oxygen saturation, ankle-brachial index (ABI), and 6-minute walking distance (6MWD) in men and women who have intermittent claudication (Fontaine Stage II; Rutherford Category 1-2) in response to 15 or 45 minutes of lower limb heating and transcutaneous electrical nerve stimulation (TENS).

ELIGIBILITY:
Inclusion Criteria:

* Intermittent claudication (Fontaine Stage II)
* Resting ankle-brachial index (ABI) < 0.90
* Ability to walk > 60 meters in six minutes

Exclusion Criteria:

* Body mass index (BMI) > 35 kg/m2
* Severe exercise limitations (more than PAD) due to co-morbidity
* Taking illegal/recreational drugs
* Uncontrolled hypertension (>180/100 mmHg)
* Severe peripheral neuropathy
* Foot ulcers
* Gangrene
* Pregnant or breast feeding

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-11-15 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Distance walked during six-minute walk test | 35 minutes post-intervention/control
  Distance walked during a self-paced six-minute walk

SECONDARY OUTCOMES:
Popliteal artery blood flow | Pre-intervention baseline; 10, 20, and 30 minutes post-intervention/control
  Unilateral popliteal blood flow measured via Doppler ultrasound
Time/distance to claudication during six-minute walk | 35 minutes following each intervention and control period
  Subjects give subjective ratings of claudication onset, if applicable, during six-minute walk test
Ankle brachial index (ABI) | Pre-intervention baseline and 20 minutes post-intervention/control
  Systolic blood pressures (SBP) are measured in the brachial arteries of both arms and in the posterior tibial and dorsalis pedis arteries of both ankles using a hand-held Doppler ultrasound probe and a sphygmomanometer
Toe oxygen saturation | Pre-intervention baseline; 10, 20, and 30 minutes post-intervention/control
  A pulse oximeter is used to measure toe oxygen saturation in the big toe of each of the subject's feet

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K. Pellinger, Ph.D., Principal Investigator — Salisbury University
Locations (1):
- Salisbury University, Salisbury, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided